CLINICAL TRIAL: NCT03204019
Title: A Phase II Randomized,Controlled,Open Label,Multicentre Study of Tegafur Combined With Temozolomide Versus Tegafur Combined With Temozolomide and Thalidomide in Subjects With Advanced Pancreatic Neuroendocrine Tumor
Brief Title: A Study of Tegafur Combined With Temozolomide Versus Tegafur Combined With Temozolomide and Thalidomide in Subjects With Advanced Pancreatic Neuroendocrine Tumor
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, yihebali chi, Assistant Professor, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CH-GI-103
Record Dates: First submitted 2017-06-28; First posted 2017-06-29 (Actual); Last update posted 2017-06-29 (Actual); Status verified 2017-06

CONDITIONS: Pancreatic Neuroendocrine Tumor
Keywords: Tegafur; Temozolomide; Thalidomide; Pancreatic Neuroendocrine Tumor
MeSH Terms: conditions — Adenoma, Islet Cell | interventions — Tegafur; Temozolomide; Thalidomide

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tegafur and Temozolomide (Experimental): Drugs should be continued until disease progression or intolerable toxicity or patients withdrawal of consent
  Interventions: Drug: Tegafur and Temozolomide
- Tegafur and Temozolomide combined with Thalidomide (Active Comparator): Drugs should be continued until disease progression or intolerable toxicity or patients withdrawal of consent
  Interventions: Drug: Tegafur and Temozolomide combined with Thalidomide

INTERVENTIONS:
Drug: Tegafur and Temozolomide — Tegafur 40-60mg po bid(d1-d14); Temozolomide 200mg po qd(d10-d14)
  Arms: Tegafur and Temozolomide
Drug: Tegafur and Temozolomide combined with Thalidomide — Tegafur 40-60mg po bid(d1-d14); Temozolomide 200mg po qe(d10-d14) Thalidomide 100mg po qd(d1-d7) /Thalidomide 200mg po qd(d8-d14)/Thalidomide 300mg po qd(d15-d21)
  Arms: Tegafur and Temozolomide combined with Thalidomide

SUMMARY:
A Phase II Randomized,Controlled,Open Label,Multicentre Study to evaluate the efficacy and safety of Tegafur combined with Temozolomide versus Tegafur combined with Temozolomide and Thalidomide in subjects with Advanced Pancreatic Neuroendocrine Tumor

ELIGIBILITY:
Inclusion Criteria:

1. Patients should participate in the study voluntarily and sign informed consent;
2. Histopathological proven diagnosis of low and intermediate grade (G1, G2 or G3) advanced pancreatic neuroendocrine tumor( locally advanced, unresectable or distant Metastatic). For gastroenteropancreatic neuroendocrine tumor（GEP-NET）,the classification is based on nuclear mitotic number and the Ki-67 index,which are as follows:G1:Nuclear mitotic number <2/10HPF,Ki-67 proliferative index ≤2%.G2: Nuclear mitotic number 2～20/10HPF,Ki-67 proliferative index 3%～20%.G3 Nuclear mitotic number >20/10HPF,Ki-67 proliferative index >20%;
3. Patients with advanced PNENs who had not been treated or had no more than two kinds of Systemic Anti-tumor Therapy,which could be somatostatin analogs, interferon, PRRT (peptide receptor radionuclide therapy), mTOR inhibitors, or chemotherapy (without any use of azole amines, fluorouracil,or thalidomide chemotherapy drugs);
4. Radiological documentation of tumor progression is required within 12 months prior to randomization;
5. At least one measurable lesion (byRECIST1.1);
6. ANC≥1.5×109/L,PLT≥100×109/L,HB≥90g/L,TBIL≤1.5ULN ;Without supportive care, ALT≤2.5ULN and ALP≤2.5ULN (without hepatic metastasis) ALT≤5ULN and ALP≤5ULN(with hepatic metastasis);serum creatin ≤1.5ULN and creatinine clearance rate ≥60ml/min；INR≤1.5ULN and APTT ≤1.5ULN ;
7. ECOG PS:0-1;
8. Life expectancy of more than 12 weeks;
9. Men/Women of childbearing potential must agree to use a highly effective contraceptive method (such as double barrier contraceptive method，condom, oral or injectable contraceptives and intrauterine device) throughout treatment and for at least 90 days after study completion；All female patients will be considered fertile unless she has undergone natural menopause, artificial menopause or sterilization (such as hysterectomy, bilateral adnexal resection, or radioactive ovarian irradiation etc.)

Exclusion Criteria:

* 1、Diagnosed with high grade (G3) neuroendocrine carcinomas, adenocarcinoma, pancreatic islet cell carcinoma, goblet cell carcinoid, large cell neuroendocrine carcinoma, and small cell carcinoma; 2、Gastrointestinal tract, lung and thymus, and other unknown source of neuroendocrine tumors; 3、Functional NET which needs concomiant use of long-acting somatostatin analogues to control symptoms such as insulinoma, gastrinoma, glucagon tumor, somatostatin, ACTH tumor, VIP tumor, and carcinoid syndrome, Zollinger-Ellison syndrome or other disease-specific active symptoms.; 4、prior use of any VEGF/VEGFR targeted drugs and with disease progression during treatment; 5、Urine protein ≥ ++，or Urine protein detected by quantitative test of 24h urinary protein>1.0 g; 6、Serum potassium and calcium (ionic or albumin binding) or magnesium exceed normal range and have clinical significance; 7、 Blood pressure unable to be stably controlled(systolic pressure>140 mmHg，diastolic pressure>90mmHg); 8、gastrointestinal diseases or states judged by Investigators that could affect the absorption of the drug, including but not limited to active gastric and duodenal ulcers, ulcerative colitis or other gastrointestinal diseases or unresectable gastrointestinal tumor with active bleeding or other status that may cause gastrointestinal bleeding or perforation; 9、Patients have or had severe hemorrhage (bleeding volume >30ml within 3 months) , hemoptysis( fresh blood >5ml within 4 weeks ) or thromboembolic events (including transient ischemic attack) within 12 months; 10、Cardiovascular disease with significant clinical significance, including but not limited to acute myocardial infarction, severe / unstable angina or coronary artery bypass surgery within 6 months prior to enrollment; congestive heart failure (New York Heart Association (NYHA) classification> 2); ventricular arrhythmia requiring pharmacological treatment; left ventricular ejection fraction (LVEF) <50%; 11、 Electrocardiogram (ECG) showed QT interval ≥480ms; 12、Patients suffered from other malignant tumors in the past 5 years,except radical resection of skin basal cells or squamous cell carcinoma, or cervical carcinoma in situ; 13、patients who have received anti-tumor therapy within 4 weeks prior to initiation of the study, including but not limited to chemotherapy, radiotherapy, bio-targeted therapy, immunotherapy, anti-tumor treatment of traditional Chinese medicine, hepatic artery embolization, hepatic metastatic cryoablation or radiofrequency ablation surgery; 14、patients who have received Palliative radiotherapy for bone metastaseswithin 2 weeks prior to initiation of the study ; 15、Any clinically significant active infection, including but not limited to HIV infection; 16、Patients with clinically significant liver disease history ,including but not limited to hepatitis B virus (HBV) infection (HBVDNA positive and copy number ≥1×104/ml); hepatitis C virus (HCV) infection,(HCVRNA positive and copy number≥1×103/ml), or cirrhosis; 17、Patients had surgery (except biopsy) within 28 days or has surgical incision not fully healed prior to initiation of the study; 18、Patients with brain metastasis or spinal cord compression which had not surgical and / or radiation therapy,or which had previous treatment but there is no clinical imaging evidence proving the condition is stable; 19、The toxic reaction of previous anticancer treatment has not restored to grade 0 or 1 (except hair loss); 20、Patients participated in other drug clinical trials within 4 weeks and received drug treatment ; 21、Pregnancy(Pregnancy test positive before drug use)or lactation; 22、any other disease, metabolic abnormality, abnormal physical examination, or laboratory abnormalities estimated by investigators that make the patients not suitable to receive the study drug or will affect the interpretation of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-10 (Actual); Primary Completion 2017-10 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate(ORR) | From randomization，each 6 weeks or 12 weeks(a year later) up to intolerance the toxicity or PD (up to 24 months)

SECONDARY OUTCOMES:
Disease Control Rate(DCR) | From randomization，each 6 weeks or 12 weeks(a year later) up to intolerance the toxicity or PD (up to 24 months
Time to Tumor Response (TTR) | From randomization，each 6 weeks or 12 weeks(a year later)up to PD or death(up to 24 months)
Duration of Response(DOR) | From randomization，each 6 weeks or 12 weeks(a year later) up to PD or death(up to 24 months)
Progression free survival(PFS) | From randomization，each 6 weeks or 12 weeks(a year later)(a year later) up to PD or death (up to 24 months)

CONTACTS AND LOCATIONS:
Overall Officials: Yihebali Chi, doctor, Principal Investigator — Chinese Academy of Medical Sciences
Locations (1):
- Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Chi Y, Song L, Liu W, Zhou Y, Miao Y, Fang W, Tan H, Shi S, Jiang H, Xu J, Jia R, Zheng B, Jiang L, Zhao J, Zhang R, Tan H, Wang Y, Chen Q, Yang M, Guo X, Tong Z, Qi Z, Zhao F, Yan X, Zhao H. S-1/temozolomide versus S-1/temozolomide plus thalidomide in advanced pancreatic and non-pancreatic neuroendocrine tumours (STEM): A randomised, open-label, multicentre phase 2 trial. EClinicalMedicine. 2022 Sep 26;54:101667. doi: 10.1016/j.eclinm.2022.101667. eCollection 2022 Dec. PMID 36188432